CLINICAL TRIAL: NCT01989286
Title: Postural Assessment in Children With Non-synostotic Plagiocephaly
Brief Title: Postural Assessment in Plagiocephaly
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Other Study IDs: DF0043UG; AP2010-3603 (Other Grant/Funding Number: Ministry of Education, Spain)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Plagiocephaly
Keywords: Plagiocephaly; Posture; Spine
MeSH Terms: conditions — Plagiocephaly | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Plagiocephaly group-Assessment: Children (3-5 years) who were diagnosed and treated because of positional plagiocephaly are included in this group. An asssessment of posture will be performed.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The posture, motor development and balance are going to be assessed.
  Other Names: Evaluation; Posture assessment; Psychomotor development

SUMMARY:
The positional plagiocephaly is a condition involving craniofacial asymmetry. The purpose of this study is to evaluate the spine, the posture and the psychomotor state in children who were diagnosed with infant plagiocephaly.

DETAILED DESCRIPTION:
Positional infant plagiocephaly is a clinical entity in which the shape of an infant's head becomes altered as the result of external forces applied to the malleable bones of the cranium and can occur pre- or postnatally. It is characterized by asymmetric occipital flattening (one side or the central part of the occiput is flattened)with ipsilateral frontal bossing.Viewed from above, this results in a parallelogram deformity of the head. We hypothesize that children who had plagiocephaly when they were infants, they have postural and spine implications at 3-5 years old.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infant positional plagiocephaly
* Aged 3, 4 or 5 years old.

Exclusion Criteria:

* Diagnosis of non synostotic plagiocephaly.
* Neurological concomitant condition.
* Problems in motor development.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who were diagnosed by plagiocephaly and a control group.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Spine assessment | baseline
  The spine alignment, segmental and global angles in the sagittal and frontal planes,and the spinal mobility are going to be assessed by the Spinal Mouse®,a device guided manually on the skin along the spine.

SECONDARY OUTCOMES:
Postural evaluation | baseline
  The postural assessment comprises the static posture and the spinal flexibility by observing different positions and actions of the children.
Psychomotor assessment | baseline
  The psychomotor development test, TEPSI, is going to be used to assess three areas: coordination, language and motor state. The children are asked to perform different activities and the success is registered.
Balance | baseline
  The balance is assessed with the Pediatric Balance Test, asking the children to perform different tasks and observing the execution of these tasks.

OTHER OUTCOMES:
Quality of sleep | baseline
  The parents are going to complete the Pediatric Sleep Questionnaire, with different items evaluating the quality of sleep of the children.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cabrera Martos, MsC, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cabrera-Martos I, Valenza MC, Valenza-Demet G, Benitez-Feliponi A, Robles-Vizcaino C, Ruiz-Extremera A. Repercussions of plagiocephaly on posture, muscle flexibility and balance in children aged 3-5 years old. J Paediatr Child Health. 2016 May;52(5):541-6. doi: 10.1111/jpc.13155. PMID 27329908